CLINICAL TRIAL: NCT03989115
Title: Ph1b/2 Open-Label,Multicenter Dose-Esc & Dose-Exp Study of Combo RMC4630 & Cobimetinib in Participants w/Relapsed/Refractory Solid Tumors & Ph1b Study of RMC4630 w/Osimertinib in Participants w/EGFR Mutation+,Locally Adv or Meta NSCLC
Brief Title: Dose-Esc/Exp RMC4630 & Cobi in Relapsed/Refractory Solid Tumors & RMC4630& Osi in EGFR+ Locally Adv/Meta NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Revolution Medicines, Inc. (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC-4630-02
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-02

CONDITIONS: Solid Tumor
Keywords: SHP2; PTPN11; NSCLC; KRAS G12; BRAF Class 3; NF1 LOF; KRAS amplification; KRAS mutations; advanced solid tumor; advanced solid malignancies; bladder cancer; carcinoma, non-small-cell lung; neoplasm, squamous cell; carcinoma, squamous cell; esophageal neoplasms carcinoma, bronchogenic; bronchial neoplasms; lung neoplasms; respiratory tract neoplasms; thoracic neoplasms; neoplasms by site; neoplasms; lung diseases; respiratory tract diseases; gastrointestinal cancer; colorectal cancer; skin cancer; ovarian cancer; pancreatic cancer; endometrium/uterus cancer; cervical cancer
MeSH Terms: conditions — Noonan Syndrome; Urinary Bladder Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms, Squamous Cell; Carcinoma, Squamous Cell; Bronchial Neoplasms; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Gastrointestinal Neoplasms; Colorectal Neoplasms; Skin Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Uterine Neoplasms; Uterine Cervical Neoplasms | interventions — cobimetinib; osimertinib

STUDY DESIGN:
Intervention Model Description: This is a dose escalation study followed by dose expansion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RMC-4630 and Cobimetinib (Experimental): RMC-4630 and Cobimetinib for oral administration
  Interventions: Drug: RMC-4630; Drug: Cobimetinib
- RMC-4630 and Osimertinib (Experimental): RMC-4630 and Osimertinib for oral administration
  Interventions: Drug: RMC-4630; Drug: Drug: Osimertinib

INTERVENTIONS:
Drug: RMC-4630 — RMC-4630 for oral administration
Drug: Cobimetinib — Cobimetinib for oral administration
  Other Names: GDC-0973, XL518
  Arms: RMC-4630 and Cobimetinib
Drug: Drug: Osimertinib — Osimertinib for oral administration
  Other Names: Tagrisso; AZD9291
  Arms: RMC-4630 and Osimertinib

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) proﬁles of RMC-4630 and cobimetinib in adult participants with relapsed/refractory solid tumors with specific genomic aberrations and to identify the recommended Phase 2 dose (RP2D); and to evaluate the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) proﬁles of RMC-4630 and osimertinib in adult participants with EGFR mutation-positive locally advanced or metastatic NSCLC.

DETAILED DESCRIPTION:
This open-label, phase 1b/2 dose-escalation and dose-expansion study is designed to evaluate the safety and maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of RMC-4630 in combination with cobimetinib in participants with relapsed/refractory solid tumors; and of RMC-4630 in combination with osimertinib in adult participants with EGFR mutation-positive locally advanced or metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* For RMC-4630 + Cobimetinib only - Participants who have advanced solid tumors that have failed, are intolerant to, or are considered ineligible for standard of care anti-cancer treatments including approved drugs for oncogenic drivers in their tumor type.
* For RMC-4630 + Osimertinib only - Locally advanced or metastatic EGFR mutant NSCLC not amenable to curative surgery or radiotherapy
* For RMC-4630 + Cobimetinib only - Participants must have one of the following genotypic aberrations: KRAS mutations and amplifications, BRAF Class 3 mutations, or NF1 LOF mutations
* For RMC-4630 + Osimertinib only - Evidence of radiological documentation of progression with osimertinib monotherapy or an osimertinib containing regimen. Participants should not be considered a current candidate for 1st generation EGFR TKI's by the investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
* Adequate hematological, hepatic, and renal function
* Capable of giving signed informed consent form (ICF). Willing and able to compile with study requirements and restrictions
* Life expectancy >12 weeks
* Female of childbearing potential and males with partners of childbearing potential must comply with effective contraception criteria .

Exclusion Criteria:

* Primary central nervous system (CNS) tumors.
* Known or suspected leptomeningeal or brain metastases or spinal cord compression.
* For RMC-4630 + osimertinib arm only - Known or suspected Small cell, squamous, or pleomorphic lung transformations
* Clinically significant cardiac disease
* Active, clinically signiﬁcant interstitial lung disease or pneumonitis
* History or current evidence of retinal pigment epithelial detachment (RPED), central serous retinopathy, retinal vein occlusion (RVO), or predisposing factors to RPED or RVO
* Known HIV infection or active/chronic hepatitis B or C infection.
* Any other unstable or clinically signiﬁcant concurrent medical condition that would, in the opinion of the investigator, jeopardize the safety of a participant, impact their expected survival through the end of the study participation, and/or impact their ability to comply with the protocol prior/concomitant therapy
* Females who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Revolution Medicines, Inc., Study Director — Revolution Medicines, Inc.
Locations (24):
- United States (21):
  - Honor Health Research Institute, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - UC Irvine - Chao Family Comprehensive Cancer Center, Orange, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Francisco - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Cancer Institute, Franz Clinic, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Dell Seton Medical Center at University of Texas, Austin, Texas
  - Virginia Cancer Specialists (Fairfax) - USOR, Fairfax, Virginia
  - University of Wisconsin, Madison, Wisconsin
- South Korea (3):
  - Severance Hospital Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center - PPDS, Seoul

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 20mg QD (21/7): Participants who received intermittent dose of RMC-4630 80 mg on D1 and D4 of a 28-day cycle and Cobimetinib 20 mg QD 21days on and 7 days off of a 28-day cycle.
- Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 40mg QD (21/7): Participants who received intermittent dose of RMC-4630 80mg on D1 and D4 of a 28-day cycle and Cobimetinib 40mg QD 21days on and 7 days off of a 28-day cycle.
- Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7): Participants who received intermittent dose of RMC-4630 140 mg on D1 and D4 of a 28-day cycle and Cobimetinib 20mg QD 21days on and 7 days off of a 28-day cycle.
- Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7): Participants who received intermittent dose of RMC-4630 140 mg on D1 and D2 of a 28-day cycle and Cobimetinib 20mg QD 21days on and 7 days off of a 28-day cycle.
- Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2): Participants who received intermittent dose of RMC-4630 140 mg on D1 and D2 of a 28-day cycle and Cobimetinib 40mg D1 and D2 of a 28-day cycle.
- Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg D1D2: Participants who received intermittent dose of RMC-4630 140 mg on D1 and D2 of a 28-day cycle and Cobimetinib 60mg D1 and D2 of a 28-day cycle.
- Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg (QD): Participants who received intermittent dose of RMC-4630 100 mg on D1 and D2 of a 28-day cycle and daily dose of Osimertinib 80 mg from D1 through D28 of a 28-day cycle.
- Intermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg (QD): Participants who received intermittent dose of RMC-4630 140 mg on D1 and D2 of a 28-day cycle and daily dose of Osimertinib 80 mg from D1 through D28 of a 28-day cycle.
Period: Overall Study
Arm/Group | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 40mg QD (21/7) | Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg D1D2 | Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg (QD) | Intermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg (QD)
Started | 8 | 6 | 12 | 7 | 65 | 7 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 6 | 12 | 7 | 65 | 7 | 4 | 4
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 0 | 17 | 1 | 0 | 0
Not completed — Sponsor decision to terminate the study | 1 | 1 | 0 | 1 | 11 | 0 | 2 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 2 | 2 | 9 | 6 | 31 | 6 | 2 | 3
Not completed — Other | 1 | 2 | 0 | 0 | 5 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 20mg QD (21/7): Participants who received intermittent dose of RMC-4630 80mg on D1 and D4 of a 28-day cycle and Cobimetinib 20 mg QD 21 days on and 7 days off of a 28-day cycle.
- Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 40mg QD (21/7): Participants who received intermittent dose of RMC-4630 80mg on D1 and D4 of a 28-day cycle and Cobimetinib 40 mg QD 21 days on and 7 days off of a 28-day cycle.
- Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7): Participants who received intermittent dose of RMC-4630 140mg on D1 and D4 of a 28-day cycle and Cobimetinib 20 mg QD 21 days on and 7 days off of a 28-day cycle.
- Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7): Participants who received intermittent dose of RMC-4630 140mg on D1 and D2 of a 28-day cycle and Cobimetinib 20 mg QD 21 days on and 7 days off of a 28-day cycle.
- Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2): Participants who received intermittent dose of RMC-4630 140mg on D1 and D2 of a 28-day cycle and Cobimetinib 40 mg D1 and D2 of a 28-day cycle.
- Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg (D1D2): Participants who received intermittent dose of RMC-4630 140mg on D1 and D2 of a 28-day cycle and Cobimetinib 60 mg D1 and D2 of a 28-day cycle.
- Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg QD: Participants who received intermittent dose of RMC-4630 100 mg on D1 and D2 of a 28-day cycle and Osimertinib 80 mg QD.
- IIntermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg QD: Participants who received intermittent dose of RMC-4630 140 mg on D1 and D2 of a 28-day cycle and Osimertinib 80 mg QD.
- Total: Total of all reporting groups
Arm/Group | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 40mg QD (21/7) | Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg (D1D2) | Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg QD | IIntermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg QD | Total
Number analyzed (Participants) | 8 | 6 | 12 | 7 | 65 | 7 | 4 | 4 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 6 | 7 | 50 | 6 | 2 | 2 | 85
  >=65 years | 0 | 2 | 6 | 0 | 15 | 1 | 2 | 2 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 5 | 2 | 34 | 4 | 2 | 2 | 58
  Male | 3 | 2 | 7 | 5 | 31 | 3 | 2 | 2 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 5 | 1 | 8 | 0 | 4 | 2 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 5
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 7 | 5 | 7 | 6 | 45 | 5 | 0 | 1 | 76
  More than one race | 0 | 0 | 0 | 0 | 7 | 2 | 0 | 0 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs).
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant, temporally associated with the use of a pharmaceutical / an investigational product, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product(s) was also an AE. All AEs and SAEs will be collected from the start of intervention until the safety visit or EOT visit, whichever is later. The number of safety-evaluable participants who experienced at least one treatment-emergent AE was reported per protocol.
Time Frame: AEs were collected from the start of intervention through 30 days post last day of study drug taken. Participants were monitored/assessed for adverse events for a maximum of 17 months which includes a maximum duration of 16 months on treatment.
Population: All safety-evaluable participants who experienced at least one treatment-emergent AE.
Measure: Count of Participants; unit: Participants
Arm/Group | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 40mg QD (21/7) | Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg D1D2 | Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg (QD) | Intermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg (QD)
Number analyzed (Participants) | 8 | 6 | 12 | 7 | 65 | 7 | 4 | 4
Participants | 8 | 6 | 12 | 7 | 64 | 7 | 4 | 4

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Any toxicities occurring during the DLT observation period (cycle 1) that were considered R/T study treatment, including GR4 AEs; GR3 febrile neutropenia or hemorrhage; GR3 thrombocytopenia with clinically significant bleeding; GR ≥2 pneumonitis; GR3 hypertension or rash which does not improve or remains uncontrolled for >5 or more days despite maximal supportive care; GR3 non hematologic AEs that remain uncontrolled for >72 hours despite maximal supportive care; Concurrent elevation of AST or ALT >3 × ULN & total bilirubin >2 × ULN or international normalized ratio (INR) >1.5 in the absence of cholestasis and other causes; Grade 3 QTcF prolongation based on a triplicate ECG; Ejection fraction <50% with an absolute decrease of >10% from baseline; Retinal vein occlusion any grade; 50% or less dose intensity of RMC4630 and/or cobimetnib or osimertinib due to study drug related toxicity. Refer to protocol for further details.
Time Frame: Cycle 1: Study Day 1 - Study Day 28 (28 days)
Population: DLT-evaluable population was defined as the following: All treated participants in the dose escalation phase who completed the DLT period and received at least 75% of planned dose of RMC-4630 and cobimetinib or RMC-4630 and Osimertinib (ie, not have missed ≥3 doses of RMC-4630 and cobimetinib on the D1D2 intermittent schedule or ≥6 doses of cobimetinib on the 21 on/7 off schedule, or ≥8 doses for reasons other than toxicity) within the DLT observation period (i.e Cycle 1)
Measure: Count of Participants; unit: Participants
Groups:
- Intermittent RMC-4630 (D1D4 or D1D2) + Daily Cobimetinib (QD21/7): Participants who received intermittent dose of RMC-4630 80 mg or 140 mg on D1 and D4 or on D1 and D2 of a 28-day cycle and daily dose of Cobimetinib 20 mg or 40 mg from D1 through D21 and then 7 days off Cobimetinib from D22 to D28 of a 28-day cycle.
- Intermittent RMC-4630 (D1D2) + Intermittent Cobimetinib (D1D2): Participants who received intermittent dose of RMC-4630 140 mg on D1 and D2 of a 28-day cycle and intermittent dose of Cobimetinib 40 mg or 60 mg on D1 and D2 of a 28-day cycle.
Arm/Group | Intermittent RMC-4630 (D1D4 or D1D2) + Daily Cobimetinib (QD21/7) | Intermittent RMC-4630 (D1D2) + Intermittent Cobimetinib (D1D2) | Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg D1D2 | Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg (QD) | Intermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg (QD)
Number analyzed (Participants) | 6 | 6 | 9 | 6 | 5 | 6 | 4 | 4
Participants | 1 | 0 | 3 | 1 | 0 | 2 | 1 | 2

3. Secondary Outcome: Cmax
Description: Peak plasma concentration of RMC-4630 and cobimetinib or RMC-4630 and osimertinib
Time Frame: 0, 0.5, 1, 2, 4, 8, 24 hours post-dose on Cycle1 Day 1 and Cycle 1 Day 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 40mg QD (21/7) | Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg D1D2 | Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg (QD) | Intermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg (QD)
Number analyzed (Participants) | 8 | 6 | 12 | 7 | 65 | 7 | 4 | 4
ng/mL
  C1D1 | 214 (45) | 248 (38) | 469 (42) | 430 (61) | 354 (52) | 449 (27) | 242 (57) | 449 (25)
  C1D15 | 207 (90) | 266 (64) | 465 (37) | 504 (71) | 395 (56) | 469 (20) | 286 (38) | 408 (3)

4. Secondary Outcome: Tmax
Description: Time to achieve peak plasma concentration of RMC-4630 and cobimetinib or RMC-4630 and osimertinib
Time Frame: 0, 0.5, 1, 2, 4, 8, 24 hours post-dose on Cycle1 Day 1 and Cycle 1 Day 15
Measure: Median (Full Range); unit: h
Arm/Group | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 40mg QD (21/7) | Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg D1D2 | Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg (QD) | Intermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg (QD)
Number analyzed (Participants) | 8 | 6 | 12 | 7 | 65 | 7 | 4 | 4
h
  C1D1 | 2.94 [1.00 to 4.13] | 2.00 [1.00 to 2.03] | 1.99 [0.90 to 7.50] | 1.02 [0.98 to 2.00] | 2.00 [0.42 to 8.00] | 1.92 [0.92 to 3.97] | 2.03 [0.98 to 7.55] | 2.95 [1.07 to 4.10]
  C1D15 | 2.04 [1.00 to 4.07] | 2.08 [0.97 to 4.99] | 3.04 [1.87 to 7.77] | 1.08 [1.00 to 2.12] | 2.00 [0.57 to 23.7] | 1.96 [0.97 to 2.07] | 1.98 [1.88 to 2.00] | 4.07 [4.05 to 4.08]

5. Secondary Outcome: Area Under the Curve (AUC)
Description: Area under the plasma concentration time curve of RMC-4630 and cobimetinib or RMC-4630 and osimertinib
Time Frame: 0, 0.5, 1, 2, 4, 8, 24 hours post-dose on Cycle1 Day 1 and Cycle 1 Day 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL x h
Arm/Group | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 40mg QD (21/7) | Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg D1D2 | Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg (QD) | Intermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg (QD)
Number analyzed (Participants) | 8 | 6 | 12 | 7 | 65 | 7 | 4 | 4
ng/mL x h
  C1D1 | 2570 (34) | 2580 (30) | 5510 (38) | 4610 (39) | 4700 (38) | 4720 (26) | 3360 (28) | 5920 (15)
  C1D15 | 3220 (91) | 3360 (44) | 6370 (37) | 5580 (45) | 5460 (45) | 5600 (18) | 4230 (35) | 5500 (26)

6. Secondary Outcome: Accumulation Ratio
Description: AUC ratio (C1D15 versus C1D1) of RMC-4630 and cobimetinib or RMC-4630 and osimertinib
Time Frame: 0, 0.5, 1, 2, 4, 8, 24 hours post-dose on Cycle1 Day 1 and Cycle 1 Day 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 40mg QD (21/7) | Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg D1D2 | Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg (QD) | Intermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg (QD)
Number analyzed (Participants) | 8 | 6 | 12 | 7 | 65 | 7 | 4 | 4
ratio | 1.36 (56) | 1.22 (24) | 1.24 (16) | 1.20 (28) | 1.19 (41) | 1.20 (41) | 1.12 (20) | 0.841 (41)

7. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response of RMC-4630 and cobimetinib or RMC-4630 and osimertinib per RECIST v1.1
Time Frame: Response assessment occurs from the start of intervention until the date of documented disease progression per RECIST 1.1 or the date of subsequent therapy, whichever occurs first.
Population: There were insufficient number of participants with events to calculate.
Measure: Median (95% Confidence Interval); unit: day(s)
Arm/Group | Intermittent RMC-4630 (D1D4 or D1D2) + Daily Cobimetinib (QD21/7) | Intermittent RMC-4630 (D1D2) + Intermittent Cobimetinib (D1D2) | Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg D1D2 | Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg (QD) | Intermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg (QD)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
day(s) |  |  |  |  | NA — insufficient number of participants with events to calculate |  |  |

8. Secondary Outcome: t1/2
Description: Elimination half-life of RMC-4630 and cobimetinib or RMC-4630 and osimertinib
Time Frame: 0, 0.5, 1, 2, 4, 8, 24 hours post-dose on Cycle1 Day 1 and Cycle 1 Day 15
Measure: Median (Full Range); unit: h
Arm/Group | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 40mg QD (21/7) | Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg D1D2 | Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg (QD) | Intermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg (QD)
Number analyzed (Participants) | 8 | 6 | 12 | 7 | 65 | 7 | 4 | 4
h
  C1D1 | 15.7 [12.3 to 20.2] | 16.1 [15.2 to 20.9] | 15.1 [11.7 to 20.6] | 16.2 [15.1 to 35.7] | 17.0 [10.8 to 26.2] | 16.9 [14.9 to 20.1] | 20.1 [14.0 to 26.2] | 16.6 [16.6 to 16.6]
  C1D15 | 20.8 [15.0 to 31.2] | 24.5 [19.8 to 29.2] | 15.7 [14.9 to 17.3] | 22.2 [16.5 to 91.7] | 14.4 [5.18 to 18.2] | 18.4 [11.3 to 24.8] | 24.6 [15.2 to 25.2] | NA [NA to NA] — Insufficient timepoints to calculate this data.

9. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the proportion of participants who achieve a CR or PR per RECIST v1.1. ORR and the corresponding 95% two-sided confidence interval were derived.
Time Frame: as for outcome 7
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 40mg QD (21/7) | Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg D1D2 | Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg (QD) | Intermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg (QD)
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 55 | 6 | 3 | 3
% of participants | 0 [0.0 to 45.9] | 0 [0.0 to 45.9] | 0 [0.0 to 36.9] | 0 [0.0 to 45.9] | 1.82 [0.0 to 9.7] | 0 [0.0 to 45.9] | 0 [0.0 to 7.1] | 0 [0.0 to 7.1]

ADVERSE EVENTS:
Time Frame: AEs were collected from the start of intervention through 30 days post last day of study drug taken. Participants were monitored/assessed for adverse events for a maximum of 17 months which includes a maximum duration of 16 months on treatment.
Description: Summary of serious treatment emergent adverse events in participants who received > / = one dose of RMC-4630 and/or cobimetinib or in all participants who received > / = one dose of RMC-4630 and/or osimertinib.
Arm/Group | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 40mg QD (21/7) | Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg D1D2 | Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg (QD) | Intermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg (QD)
All-Cause Mortality (participants affected / at risk) | 2/8 | 2/6 | 9/12 | 6/7 | 31/65 | 6/7 | 2/4 | 3/4
Serious Adverse Events (participants affected / at risk) | 2/8 | 4/6 | 3/12 | 3/7 | 29/65 | 3/7 | 1/4 | 1/4
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6 | 12/12 | 7/7 | 64/65 | 7/7 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 20mg QD (21/7) (N=8) | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 40mg QD (21/7) (N=6) | Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7) (N=12) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7) (N=7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2) (N=65) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg D1D2 (N=7) | Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg (QD) (N=4) | Intermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg (QD) (N=4)
gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 (0)
large intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 0
sepsis (Infections and infestations) | 0 (0) | 0 | 1 | 0 | 2 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0
haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 (0) | 0 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
myocardial infarction (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 20mg QD (21/7) (N=8) | Intermittent RMC-4630 80mg (D1D4) + Cobimetinib 40mg QD (21/7) (N=6) | Intermittent RMC-4630 140mg (D1D4) + Cobimetinib 20mg QD (21/7) (N=12) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 20mg QD (21/7) (N=7) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 40mg (D1D2) (N=65) | Intermittent RMC-4630 140mg (D1D2) + Cobimetinib 60mg D1D2 (N=7) | Intermittent RMC-4630 100mg (D1D2) + Osimertinib 80mg (QD) (N=4) | Intermittent RMC-4630 140mg (D1D2) + Osimertinib 80mg (QD) (N=4)
diarrhoea (Gastrointestinal disorders) | 6 | 6 | 11 | 6 | 53 | 7 | 3 | 4
nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 1 | 24 | 3 | 0 | 0
constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 19 | 1 | 0 | 1
vomiting (Gastrointestinal disorders) | 2 | 2 | 2 | 1 | 13 | 3 | 0 | 1
abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2 | 2 | 14 | 1 | 1 | 0
abdominal distention (Gastrointestinal disorders) | 2 | 3 | 1 | 1 | 9 | 2 | 0 | 0
dry mouth (Gastrointestinal disorders) | 2 | 1 | 2 | 2 | 9 | 0 | 0 | 1
ascites (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 4 | 0 | 0 | 0
fatigue (General disorders) | 1 | 3 | 3 | 3 | 23 | 2 | 4 | 1
oedema peripheral (General disorders) | 2 | 2 | 4 | 1 | 22 | 1 | 0 | 1
pyrexia (General disorders) | 1 | 1 | 3 | 1 | 13 | 1 | 0 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 5 | 2 | 21 | 1 | 2 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 9 | 0 | 1 | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1 | 7 | 0 | 2 | 0
aspartate aminotransferase increased (Investigations) | 1 | 2 | 2 | 4 | 11 | 0 | 0 | 0
platelet count decreased (Investigations) | 1 | 1 | 2 | 2 | 10 | 0 | 1 | 1
blood creatine phosphokinase increased (Investigations) | 0 | 3 | 2 | 2 | 6 | 2 | 0 | 0
lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 5 | 1 | 1
decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 14 | 0 | 0 | 3
hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 11 | 1 | 0 | 1
hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 1 | 5 | 1 | 1 | 0
dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 7 | 2 | 1 | 2
hyponatraemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 1 | 5 | 0 | 0 | 1
anaemia (Blood and lymphatic system disorders) | 1 | 3 | 5 | 4 | 23 | 1 | 1 | 1
thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 2 | 7 | 2 | 0 | 1
vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 10 | 1 | 0 | 0
rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1 | 4 | 0 | 2 | 0
dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 4 | 0 | 2 | 0
dizziness (Nervous system disorders) | 2 | 1 | 2 | 2 | 11 | 0 | 0 | 2
fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1
gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
reticulocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
scrotal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0
asthenia (General disorders) | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0
chills (General disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0
face oedema (General disorders) | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0
peripheral swelling (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
generalised oedema (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
localised oedema (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
oedema (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 10 | 0 | 1 | 0
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
blood alkaline phosphatase increased (Investigations) | 0 | 2 | 1 | 1 | 6 | 0 | 0 | 0
weight increased (Investigations) | 1 | 0 | 2 | 0 | 7 | 0 | 0 | 0
blood creatinine increased (Investigations) | 2 | 1 | 0 | 0 | 6 | 0 | 1 | 0
gamma-glutamyltranferase increased (Investigations) | 0 | 0 | 0 | 1 | 5 | 1 | 0 | 0
alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0
blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 4 (4) | 0 | 0 | 0 (0)
white blood cell count decreased (Investigations) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 12 | 1 | 1 | 0
weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 1
dry eye (Eye disorders) | 1 | 0 | 2 | 0 | 3 | 0 | 0 | 0
dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 5 | 2 | 0 | 1
rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 4 | 1 | 0 | 0
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 6 | 0 | 0 | 0
syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 4 | 1 | 0 | 0
pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 6 | 0 | 0 | 0
haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 4 | 0 | 0 | 0
hypotension (Vascular disorders) | 0 | 1 | 2 | 1 | 6 | 2 | 0 | 0
hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 7 | 0 | 3 | 0
leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
periorbital oedema (Eye disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 7 | 0 | 0 | 0
abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
hernia (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
swelling face (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0
haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ejection fraction decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
blood uric acid decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
blood uric acid increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
international normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
protein total decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
troponin T increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
troponin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0
hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
hypouricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
retinopathy (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
subretinal fluid (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 20 | 1 | 0 | 0
chorioretinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
detachment of retinal pigment epithelium (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
palmer-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
hypoaesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
taste disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
rash pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
onychomycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0
depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
anisomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT03989115/Prot_SAP_000.pdf